CLINICAL TRIAL: NCT06896084
Title: Comparison of Surgeons' Object Discernment Via Their Hands Versus Using a Robotic Surgical System That Does Not Incorporate Haptics
Status: Completed | Type: Observational
Sponsor: Valley Health System (Other)
Responsible Party: Sponsor
Other Study IDs: II_Culligan_24JUN23
Record Dates: First submitted 2024-08-19; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Health Services Research

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Group A: Board Certified Surgeons
  Interventions: Device: da Vinci Xi System
- Group B: Robotic Board Certified Surgeons
  Interventions: Device: da Vinci Xi System

INTERVENTIONS:
Device: da Vinci Xi System — A group of surgeons will make determinations as to the material within identical balloons while using the da Vinci Xi System

SUMMARY:
The purpose of this study is to compare surgeons' discernment of 4 balloons filled with different materials when using their eyes and hands versus using the da Vinci robot.

DETAILED DESCRIPTION:
The study design is a non-randomized parallel group study in which a group of surgeons (Group A) will make determinations as to the material within each of four visually identical balloons that contain air, water, petroleum jelly or a firm substance similar to the consistency of a non-ripe banana using their hands and eyes while another group of experienced robotic surgeons (Group B) will do so using the da Vinci Xi System (Intuitive Surgical, Sunnyvale, CA).

Before making their "hands on" determinations as to balloon contents, each participant will be asked to first determine whether they can visually determine the balloon contents without any manipulation. For the purposes of outcome measurement, only two possible outcomes are considered - namely that the 4 balloons are ordered correctly or not.

Investigators will also record each "guess" for all participants in order to report any trends of mis-assortment that may occur.

ELIGIBILITY:
Inclusion Criteria:

* Board Certified Surgeon
* Robotic Board Certified Surgeon

Exclusion Criteria:

• Non Board Certified Surgeon

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Targeted population are board certifed surgeons and those who are robotic certified surgeons
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-08-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with Farrington-Manning test of Binary Non-Inferiority | 1 month
  Using the Farrington-Manning test of binary non-inferiority, investigators hypothesize that 100% correct balloon discernment by hands-on surgeons and prospectively set 80% correct discernment by robotic surgeons as their definition of non-inferiority. A correct response is a binary outcome for each of the four balloons.

CONTACTS AND LOCATIONS:
Locations (1):
- The Valley Hospital, Ridgewood, New Jersey, United States

DOCUMENTS (1):
  • Study Protocol (2023-06-24): https://cdn.clinicaltrials.gov/large-docs/84/NCT06896084/Prot_000.pdf